CLINICAL TRIAL: NCT06277791
Title: A Single Arm, Exploratory Clinical Study of the Combination of Adebrelimab and TP Regimen for Neoadjuvant Therapy in Patients With Stage IVB Oral Squamous Cell Carcinoma in Clinical Practice
Brief Title: The Combination of Adebrelimab and TP Regimen for Neoadjuvant Therapy in Patients With Stage IVB Oral Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital of Stomatology, Wuhan University (Other)
Responsible Party: Principal Investigator, Jun Jia, Associate Professor, Hospital of Stomatology, Wuhan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HStomatologyWuhan1
Record Dates: First submitted 2024-01-30; First posted 2024-02-26 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Clinical IVb Stage Oral Squamous Cell Carcinomas Patients
Keywords: Adebrelimab; PD-L1; Neoadjuvant therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): TP: docetaxel 75 mg/m2, cisplatin 75 mg/m2 Adebrelimab: 20mg/kg, intravenous infusion, D1 Every three weeks, a total of two cycles. Surgery will be performed 1-3 weeks after the completion of neoadjuvant therapy.
  After surgery, radiotherapy and chemotherapy combined with immunotherapy were chosen based on the patient's condition, and a total of two years of follow-up were conducted.
  Interventions: Drug: Adebrelimab

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab：20mg/kg, ivdrip, D1，Q3W

SUMMARY:
The goal of this [type of study:clinical trial] is to [learn about] in [Clinical IVB stage oral squamous cell carcinoma patients]. The main question it aims to answer are:

• [Observing the effectiveness and safety of the combination of Adebrelimab and TP regimen in neoadjuvant therapy for clinical IVB stage oral squamous cell carcinoma patients] Participants will [Received treatment with Adebrelimab combined with TP regimen, followed by surgery after 2 cycles of neoadjuvant therapy. After surgery, radiotherapy and chemotherapy combined with immunotherapy were chosen based on the patient's condition, with a total follow-up of two years.].

ELIGIBILITY:
Inclusion Criteria:

1. Oral squamous cell carcinoma patients diagnosed by histology or cytology;
2. Has not received any treatment for oral squamous cell carcinoma in the past;
3. According to the AJCC TNM staging system, stage clinical IVB;
4. ECOG score: 0-1 points;
5. Expected survival time ≥ 12 weeks;
6. The main organ function is good, and the laboratory test data meets the following standards: (1) Blood routine: Absolute neutrophil count ≥ 1.5 × 109/L (or greater than the lower limit of normal values in the research center laboratory), platelet count ≥ 100 × 109/L, hemoglobin ≥ 90g/L; (2) Liver function: serum total bilirubin ≤ 1.5 times the upper limit of the standard value (ULN), AST and ALT ≤ 2.5 times the ULN. If the patient has liver metastasis, this standard is ≤ 5 times the ULN; (3) Renal function: CrCl ≥ 60 ml/min/1.73 m2 (calculated according to Cockcroft Gault formula);
7. Female participants with fertility, as well as male participants with partners who are fertile women, are required to use a medically recognized contraceptive measure (such as an intrauterine device, contraceptive pill, or condom) during the study treatment period, and at least 6 months after the last use of adelbizumab and at least 6 months after the last use of chemotherapy;
8. Voluntarily participate in this study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. There are uncontrollable pleural effusion, pericardial effusion, or abdominal effusion that require repeated drainage;
2. Have a history of allergies to any components of adelbizumab in the past;
3. Have received any of the following treatments:

   1. Received any other investigational medication within 4 weeks prior to the first use of the investigational medication, or had a half-life of no more than 5 weeks from the last investigational medication;
   2. Simultaneously enroll in another clinical study, unless it is an observational (non intervention) clinical study or an intervention clinical study follow-up;
   3. Received anti-tumor therapy (including radiotherapy, chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biological therapy, or tumor embolization) within 2 weeks prior to the first use of the investigational drug;
   4. Subjects who need to receive corticosteroids (>10mg prednisone equivalent dose per day) within 2 weeks prior to the first use of the study drug. Allow the use of hormones for routine chemotherapy pretreatment without the need for dose adjustment. Other special circumstances require communication with the researcher. In the absence of active autoimmune diseases, it is allowed to inhale or locally use steroids and adrenal cortex hormone replacement with a dose greater than 10mg/day of prednisone efficacy dose;
   5. Individuals who have received anti-tumor vaccines or have received live vaccines within 4 weeks prior to the first administration of the investigational drug;
   6. Having undergone major surgery or severe trauma within 4 weeks prior to the first use of the investigational drug;
   7. Patients who have previously received treatment with paclitaxel drugs;
4. The toxicity of previous anti-tumor treatments has not recovered to ≤ CTCAE 5.0 level 1 (excluding hair loss) or the level specified by the inclusion/exclusion criteria;
5. A history of active autoimmune diseases and autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to the above diseases or syndromes); Excluding patients with vitiligo or childhood asthma/allergies who have already recovered and do not require any intervention in adulthood; Autoimmune mediated hypothyroidism treated with stable doses of thyroid replacement hormone; Type I diabetes with a stable dose of insulin;
6. Have a history of immune deficiency, including HIV test positive, or have other acquired or congenital immune deficiency diseases, or have a history of organ transplantation and allogeneic bone marrow transplantation, or active hepatitis (hepatitis B reference: HBV DNA test value exceeds 500 IU/ml or 2500 copies/mL);
7. The subjects have uncontrolled cardiovascular clinical symptoms or diseases, including but not limited to: (1) NYHA grade II or above heart failure; (2) Unstable angina pectoris; (3) Have experienced myocardial infarction within one year; (4) Clinically significant supraventricular or ventricular arrhythmias that have not been clinically intervened or are still poorly controlled after clinical intervention;
8. Serious infections (CTCAE 5.0>Level 2) occurred within 4 weeks prior to the first use of the study drug, such as severe pneumonia, bacteremia, and infection complications that require hospitalization treatment; Baseline chest imaging examination suggests the presence of active pulmonary inflammation, symptoms and signs of infection within 2 weeks prior to the first use of the study drug, or the need for oral or intravenous antibiotic treatment, excluding prophylactic use of antibiotics;
9. History of interstitial lung disease (excluding radiation pneumonia and non infectious pneumonia that have not been treated with steroids);
10. Patients who have been diagnosed with active pulmonary tuberculosis infection through medical history or CT examination, or have a history of active pulmonary tuberculosis infection within one year before enrollment, or have a history of active pulmonary tuberculosis infection more than one year before but have not received formal treatment;
11. Diagnosed with any other malignant tumor within the 5 years prior to the first use of the investigational drug, excluding malignant tumors with low risk of metastasis and mortality (5-year survival rate>90%), such as basal cell or squamous cell skin cancer or cervical carcinoma in situ that has been adequately treated;
12. Pregnant or lactating women;
13. According to the researcher's judgment, there are other factors that may cause the subject to be forced to terminate the study midway, such as other serious illnesses (including mental illness) requiring concurrent treatment, severe abnormalities in laboratory test values, family or social factors, which may affect the safety of the subject or the collection of trial data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-08-19 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Effective mitigation rate（EMR） | From enrollment to the end of surgery,assessed up to 6 months
  Pathological complete remission（PCR）+Major pathological relief（MPR）

SECONDARY OUTCOMES:
DFS | From enrollment to the first appearance of disease progression or date of death from any cause,whichever came first, assessed up to 36 months
  Disease free survival
R0 resection rate | From enrollment to the end of surgery,whichever came first, assessed up to 6 months
  :R0 is the ratio of no residue under the microscope after resection
ORR | From enrollment to initial efficacy evaluation,assessed up to 6 months
  Objective response rate
mOS | From enrollment to patient death,assessed up to 50 months
  Median overall survival

CONTACTS AND LOCATIONS:
Overall Officials: J Jia, Associate Professor, Study Director — School of Stomatology Wuhan University
Locations (1):
- School of Stomatology Wuhan University, Hubei, Wuhan, China

IPD SHARING:
Plan to Share IPD: No